CLINICAL TRIAL: NCT02596867
Title: Pilot "Window of Opportunity" Neoadjuvant Study of Propranolol in Breast Cancer
Brief Title: Neoadjuvant Propanolol in Breast Cancer
Acronym: NPBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Zeina Nahleh, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E15123
Record Dates: First submitted 2015-09-02; First posted 2015-11-04 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: B adrenergic pathway; B Blocker
MeSH Terms: conditions — Breast Neoplasms | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label single arm, drug propanolol (Experimental): all subjects will receive the experimental drug
  Interventions: Drug: propanolol

INTERVENTIONS:
Drug: propanolol — Participants will take 1.5 mg/kg/day propranolol, twice daily for 3 weeks until surgical resection of the breast tumor is performed

SUMMARY:
This trial is a Phase II study using the "window-of-opportunity" design in which the treatment-free window between breast cancer diagnosis and surgical tumor resection is used to study the biological effects of the beta blocker propranolol .

DETAILED DESCRIPTION:
* Patients will be recruited from the Garbar Breast Care Center and University Medical Center following diagnosis of invasive breast cancer by breast biopsy.
* The sympatholytic nonselective beta blocker propranolol will be administered to all participants in a non-randomized manner at an equal dose of 1.5 mg/kg/day.
* Following surgical resection of the tumor , the primary endpoint of this study is quantified by comparing the proliferative index of the tumor before propranolol administration (quantified using the initial tumor biopsy) and after 3 weeks of propranolol (quantified using the surgically resected tumor).
* Additional molecular analyses and evaluation of safety and toxicity will also be performed to better understand the effects of this treatment on breast cancers and patient adherence to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18- 65
* diagnosis of stage I-III breast cancer , confirmed by a core biopsy
* Planning to undergo definitive surgery including mastectomy or breast conserving surgery
* Systolic blood pressure must be >100 mmHg but no more than 140 mmHg and/or diastolic > 60 mmHg and no more than 95 mmHg.
* normal baseline EKG

Exclusion criteria:

* Pregnancy; potential subjects of female bearing age will have to complete a pregnancy test during screening to ensure that they are not pregnant. Potential patients who are post-menopausal must have confirmed one year without menstrual cycle.
* Free of major medical illnesses including:
* Uncontrolled Diabetes (HbA1c of ≤ 8 if previously tested)
* Uncontrolled hypertension: BP >systolic 140/ diastolic > 95
* Cardiac diseases (history of cardiac valve disease, coronary artery disease, congestive heart failure, A-V block, peripheral vascular disease, any cardiac arrhythmia/bradycardia) with the exception of the diagnosed cancer.
* Histories of asthma, bronchospastic disease, or obstructive pulmonary disease
* Previously diagnosed thyrotoxicosis
* Severe allergic reactions to medications which are included in the beta blocker family
* Previously or currently treated with a beta adrenergic receptor antagonist
* Patients with locally advanced or inflammatory breast cancer not amenable to surgical resection
* Patients taking any of the following medications will be excluded:

  * Drugs that are categorized as digitalis glycosides, beta-blockers and calcium channel blockers, ACE inhibitors and alpha blockers
  * Amiodarone
  * Cimetidine
  * Ciprofloxacin
  * Delavudin
  * Dobutamine
  * Ethanol
  * Fluconazole
  * Fluoxetine
  * Fluvoxamine
  * Haloperidol
  * Imipramine
  * Isoniazid
  * Isoproterenol
  * Luvoxamine
  * Paroxetine
  * Phenytoin
  * Phenobarbital.
  * Propafenone.
  * Quinidine
  * Reserpine
  * Rifampin
  * Ritonavir
  * Rizatriptan.
  * Tenioposide
  * Theophylline
  * Thyroxine
  * Tolbutamide.
  * Warfarin
  * Zileuton
  * Zolmitriptan

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University HSC, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
if the study is completed, yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective - two breast cancer patients enrolled over 6 months perios from clinic .
Groups:
- Open Label Single Arm, Drug Propanolol: 2 subjects enrolled and received the experimental drug propanolol: Participants took 1.5 mg/kg/day propranolol, twice daily for 3 weeks until surgical resection of the breast tumor is performed
Period: Overall Study
Arm/Group | Open Label Single Arm, Drug Propanolol
Started | 2
2 Patients Prospectively Recruited | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Single Arm, Drug Propanolol
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Tumor response by Ki 67 [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effect of the Beta Blocker Propranolol on Reducing the Tumor Proliferative Index Using Ki-67.
Description: to evaluate effect of beta adrenergic blockades on breast cancer at by Ki67 percentage change- we are looking at at least 10% mean change in the tumor proliferative index following propranolol treatment
Time Frame: 3 weeks
Population: Two patients with breast cancer are included in this analysis. One patient was a stage I breast cancer and the second patient was a stage III breast cancer.
Measure: Number; unit: % mean difference of Ki67
Groups:
- Open Label Single Arm, Drug Propanolol: We tested the efficacy of propranolol on two patients with breast cancer by recording % reduction of Ki67
Arm/Group | Open Label Single Arm, Drug Propanolol
Number analyzed (Participants) | 2
% mean difference of Ki67
  Stage I Patient 1: number analyzed (Participants) | 1
  Stage I Patient 1 | 23
  Stage III Patient 2: number analyzed (Participants) | 1
  Stage III Patient 2 | 66

2. Secondary Outcome: Assess the Safety, Toxicity and Adherence to Propranolol.
Description: Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.(Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4)
Time Frame: 3 weeks
Population: Two patients with breast cancer are included in this analysis. One patient was a stage I breast cancer and the second patient was a stage III breast cancer, AEs were assessed during and after treatment
Measure: Count of Participants; unit: Participants
Groups:
- Open Label Single Arm, Drug Propanolol: 2 subjects enrolled and received the experimental drug
  propanolol: Participants took 1.5 mg/kg/day propranolol, twice daily for 3 weeks until surgical resection of the breast tumor is performed
  Both patients reported no AEs due to treatment during treatment phase
Arm/Group | Open Label Single Arm, Drug Propanolol
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: AEs were monitored during and at the end of treatment (a total of 3 weeks)
Description: Zero AEs were reported/observed during and at the end of treatment. Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4
Arm/Group | Open Label Single Arm, Drug Propanolol
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
slow accrual was noted , mostly due to scheduling of surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02596867/Prot_SAP_000.pdf